CLINICAL TRIAL: NCT06968026
Title: Effects of High-Intensity, Low-Frequency Periodic rTMS Over the Right Dorsolateral Prefrontal Cortex on Cardiac Autonomic Regulation in Women With Recurrent Pregnancy Loss and Anxiety: A Proof-of-Concept rTMS-ECG Clinical Trial ( NEURO-CARD)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shenyang Jinghua Hospital (Industry)
Collaborators: Central Hospital Affiliated to Shenyang Medical Collage (Other); Shenyang Medical College (Other); The Second Hospital of Shenyang Medical College (Other); 242 Hospital Affiliated to Shenyang Medical College (Unknown)
Responsible Party: Principal Investigator, Lin Tao, Assoc. Prof., Shenyang Medical College
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0413
Record Dates: First submitted 2025-05-03; First posted 2025-05-13 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Recurrent Pregnancy Loss; Anxiety Disorders
Keywords: Recurrent pregnancy loss; anxiety disorders; repetitive transcranial magnetic stimulation; dorsolateral prefrontal cortex; autonomic modulation
MeSH Terms: conditions — Anxiety Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: This study adopts a sequential interventional model in which all participants receive a single-arm intervention consisting of six consecutive stimulation blocks of low-frequency rTMS targeting the right dorsolateral prefrontal cortex (DLPFC). Each participant undergoes stimulation at increasing intensities (100% to 150% of resting motor threshold [RMT]) in a fixed, predefined sequence. The design allows for within-subject comparisons across stimulation intensities, with no randomization or crossover between different intervention arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- rTMS Intervention (Experimental): This study is designed as a proof-of-concept clinical trial, employing a within-subject, single-factor repeated-measures design
  Interventions: Device: repetitive transcranial magnetic stimulation(rTMS)

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation(rTMS) — The eligible participants will undergo an intensity sweep consisting of six stimulation trains over the right dorsolateral prefrontal cortex (DLPFC), with stimulation intensities ranging from 100% to 150% of the individual resting motor threshold (RMT), increasing in 10% increments. Each train will last 60 seconds, comprising 40 seconds of active rTMS at 1 Hz and a 20-second intertrain interval (ITI). Synchronous electrocardiogram (ECG) data will be continuously recorded throughout the entire procedure.

SUMMARY:
This proof-of-concept trial investigates whether high-intensity, low-frequency repetitive transcranial magnetic stimulation (rTMS) targeting the right dorsolateral prefrontal cortex (DLPFC) can improve autonomic cardiac regulation in women with recurrent pregnancy loss (RPL) and anxiety. The study explores the lateralised function of the DLPFC in emotional and autonomic control and tests a novel neuromodulation-based strategy to relieve anxiety and sympathetic overactivation.

DETAILED DESCRIPTION:
Recurrent pregnancy loss (RPL) is frequently associated with persistent anxiety and cardiac autonomic dysregulation, forming a vicious cycle that impacts emotional and reproductive outcomes. Neuroimaging studies suggest that lateralised dysfunction of the dorsolateral prefrontal cortex (DLPFC) contributes to both emotional dysregulation and sympathetic overactivation.

Building upon the proposed Brain-Heart-Emotion interaction model, we hypothesise that excessive right DLPFC activity amplifies emotional arousal and cardiac sympathetic drive, while insufficient left DLPFC regulation fails to provide cognitive control over anxiety. This imbalance may underlie the comorbidity of anxiety and autonomic dysfunction in women with RPL.

This proof-of-concept clinical trial applies high-intensity, low-frequency repetitive transcranial magnetic stimulation (rTMS) to the right DLPFC, aiming to assess its acute neurocardiac effects, specifically rTMS-induced changes in heart rate and heart rate variability (HRV)-two key indicators of autonomic modulation.

By using a sequential stimulation paradigm combined with real-time ECG acquisition, this trial will identify the optimal intensity threshold for autonomic modulation and determine whether right DLPFC-targeted rTMS can transiently reduce cardiac sympathetic tone.

Findings from this study will inform future trials evaluating rTMS as a precision treatment for anxiety and autonomic dysfunction in RPL, potentially improving psychophysiological health and pregnancy outcomes without relying on pharmacotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Female, aged 18-45 years, and right-handed.
2. Diagnosis of recurrent pregnancy loss (RPL), defined as ≥2 consecutive spontaneous miscarriages before 28 weeks of gestation.
3. Currently non-pregnant, or presenting with a missed abortion (no fetal cardiac activity confirmed by ultrasound).
4. Hamilton Anxiety Rating Scale (HAMA) score ≥14 (moderate or greater anxiety) and Hamilton Depression Rating Scale (HAMD-17) score ≤17 (to exclude clinically significant depression).
5. Confirmed diagnosis of at least one DSM-5 anxiety disorder subtype-generalized anxiety disorder (GAD), panic disorder (PD), social anxiety disorder (SAD), or post-traumatic stress disorder (PTSD)-based on a structured or semi-structured psychiatric interview conducted remotely via HIPAA-compliant, encrypted video by a board-certified psychiatrist.--Exclusion Criteria:

1) Contraindications to transcranial magnetic stimulation (TMS), including metallic implants or a history of epilepsy; 2) Uncontrolled blood pressure (systolic >180 mmHg or <90 mmHg); 3) Presence of other major medical conditions, including hyperthyroidism, a history of atrial fibrillation, valvular heart disease, sinus bradycardia, neurological disorders, cerebrovascular disease, or chronic pulmonary disease; 4) Clinically significant suicide risk; 5) A current or past diagnosis of other psychiatric disorders, including substance use disorders, schizophrenia, delusional disorder, unspecified psychotic disorder, bipolar disorder, or delirium.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women with recurrent pregnancy loss and anxiety
Enrollment: 55 (Estimated)
Dates: Start 2025-05-16 (Actual); Primary Completion 2026-03-13 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Change in baseline-corrected heart rate across stimulation intensities | During six consecutive stimulation trains (each 60 seconds; intensities increasing from 100% to 150% RMT)
  Mean baseline-corrected heart rate will be calculated for each stimulation intensity to assess autonomic cardiac responses to increasing low-frequency rTMS intensity
Change in heart rate variability (HRV) spectral power at 0.0167 Hz during rTMS | During six consecutive stimulation trains (each 60 seconds; intensities increasing from 100% to 150% RMT
  HRV spectral power at the entrainment frequency (0.0167 Hz) will be extracted from ECG data and compared across stimulation intensities to assess rhythmic autonomic modulation

SECONDARY OUTCOMES:
Brain-Heart Coupling (BHC) strength at each stimulation intensity | During six consecutive stimulation trains (100% to 150% RMT)
  BHC will be calculated as the Pearson correlation between stimulation-induced changes in heart rate and frequency-specific HRV power (at 0.0167 Hz) within the stimulation window
Incidence of non-serious adverse events | Immediately after the rTMS session
  Participants will be monitored for stimulation-site discomfort, transient facial muscle twitching, mild headache, or dizziness
Incidence of serious adverse events | Immediately after the rTMS session
  Serious adverse events, including syncope or seizure, will be recorded if they occur following the rTMS procedure

CONTACTS AND LOCATIONS:
Overall Officials: Lin Tao, MM, Principal Investigator — Shenyang Medical College; Yun-En Liu, MD, Study Chair — Shenyang Medical College
Locations (3):
- China (3):
  - The Second Affiliated Hospital of Shenyang Medical College, Shenyang, Liaoning
  - Shenyang Jinghua Hospital, Shenyang, Liaoning
  - Central Hospital Affiliated to Shenyang Medical Collage, Shenyang, Liaoning

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data, along with the study protocol, analysis scripts, and supporting materials, will be made available at the time of publication of the final article. Data will be deposited on the ResMan platform (http://www.medresman.org.cn/) and will be accessible for non-commercial research purposes. Requests for additional materials or clarifications may be directed to the corresponding author.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Available at the time of publication of the final article
Access Criteria: Data will be deposited on the ResMan platform and will be accessible for non-commercial research purposes.